CLINICAL TRIAL: NCT00467298
Title: An Intervention to Enhance Function in Severe Cardiopulmonary Illness
Brief Title: An Intervention to Improve Function in Severe Cardiopulmonary Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NRI 04-242
Record Dates: First submitted 2007-04-25; First posted 2007-04-30 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Heart Failure
Keywords: Exercise; heart failure; chronic obstructive pulmonary disease; patient education; costs; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-management (Experimental): Novel intensive self-management education and exercise program of four weeks
  Interventions: Behavioral: Exercise adherence; Behavioral: Self-management- prevention of illness; Behavioral: Self-management of illness
- Usual care (No Intervention): Usual care- cardiac or pulmonary rehabilitation exercise program of 8 weeks duration

INTERVENTIONS:
Behavioral: Exercise adherence — The exercise program includes endurance and strength training and warm-up and cool-down strategies. Emphasis is placed upon implementing and adhering to the exercise program at home following intervention completion.
  Arms: Self-management
Behavioral: Self-management- prevention of illness — Instruction is provided regarding key elements of managing heart failure and COPD with emphasis upon individual adaptations to prevent exacerbations, unscheduled provider visits, and hospital admissions as well as promotion of daily activity.
  Arms: Self-management
Behavioral: Self-management of illness — This component of the intervention stresses the use of an action plan that is implemented to c-manage bouts of mild illness and to identify symptoms of more serious illness, including appropriate actions.
  Arms: Self-management

SUMMARY:
The study is a randomized trial of a cardiopulmonary self-management intervention to improve functional capacity, health-related quality of life, and to reduce health care utilization. Two hundred (100 in each group) will be recruited from VA Puget Sound Health Care System over four years. Outcomes will be measured at three points: at entry, at the end of the 6 month intervention, and 12 months after entry. Change in functional capacity at the end of the intervention program is the primary outcome.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial of a cardiopulmonary exercise and self-management intervention to improve functional capacity, health related-related quality of life, and to reduce health care costs in medically fragile, elderly patients with chronic obstructive pulmonary disease (COPD) or heart failure (HF). Specific aims include: (1) To determine the benefits of a combined outpatient/home-based exercise, self-management program on function al capability (daily activity, six-minute walk distance, symptoms), (2) to determine the effects of exercise/self-management on quality of life, health status, cardiopulmonary function, and gait and balance, (3) to test the theoretical self-regulation model for mediating effects on major outcome variables, and (4) to compare health care resource utilization and expenditures between the intervention and usual care groups in order to conduct a cost-effectiveness analysis of the program. The primary outcome upon which the study is powered is functional capability measured by daily physical activity. Outcomes will be measured at three time points: at entry and following the intervention at 6 and 12 months. Two-hundred (100/group) will be recruited from the VA Puget Sound Health Care System outpatient clinics. The study will be carried out over four years. Inclusion criteria include standard criteria for severe COPD or HF, optimal medical management, willingness to participate in an outpatient exercise/self-management program, working phone, hospitalization for HF, COPD, or related illness in the past two years or at least two outpatient visits for same over the past year. Exclusion criteria include unstable disease or recent surgery, supplemental oxygen requirement at rest more than 4 LPM, already participating in regular exercise three times a week, inability to ambulate, uncontrolled mental illness, alcohol or drug abuse and life expectancy less than one year. The intervention consists of a month long program of two 2-hour visits a week incorporating equal time for endurance and strength training as well as individually-tailored instruction in self-management of their heart/lung disease. Usual care control is an 8-week standard cardiopulmonary exercise program, two days a week for an hour with some self-management content.

ELIGIBILITY:
Inclusion Criteria:

* standard criteria for severe COPD or HF,
* optimal medical management,
* willingness to participate in an outpatient exercise/self-management program,
* working phone,
* hospitalization for HF, COPD, or related illness in the past two years or at least two unscheduled outpatient visits for same over the past year

Exclusion Criteria:

* unstable disease or recent surgery,
* supplemental oxygen requirement at rest more than 4 LPM,
* already participating in regular exercise three times a week,
* inability to ambulate,
* uncontrolled mental illness,
* alcohol or drug abuse,
* life expectancy less than one year

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie G. Steele, PhD RN, Principal Investigator — VA Puget Sound Health Care System; Cynthia M. Dougherty, PhD RN, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Steele BG, Belza B, Cain KC, Coppersmith J, Lakshminarayan S, Howard J, Haselkorn JK. A randomized clinical trial of an activity and exercise adherence intervention in chronic pulmonary disease. Arch Phys Med Rehabil. 2008 Mar;89(3):404-12. doi: 10.1016/j.apmr.2007.11.003. PMID 18295615
- [Background] Steele BG, Cain K, Coppersmith J, Belza B, Howard J, Lakshminarayan S. Pulmonary rehabilitation (PR) outcomes in chronic obstructive pulmonary disease (COPD): Are benefits equivalent in end-stage disease? Proceedings of the American Thoracic Society. 2008 May 17; 177:A446.
- [Background] Steele BG, Belza B, Cain K, Coppersmith J, Howard J, Lakshminarayan S, Haselkorn J. The impact of chronic obstructive pulmonary disease exacerbation on pulmonary rehabilitation participation and functional outcomes. J Cardiopulm Rehabil Prev. 2010 Jan-Feb;30(1):53-60. doi: 10.1097/HCR.0b013e3181c85845. PMID 20068424
- [Result] Nguyen HQ, Gill DP, Wolpin S, Steele BG, Benditt JO. Pilot study of a cell phone-based exercise persistence intervention post-rehabilitation for COPD. Int J Chron Obstruct Pulmon Dis. 2009;4:301-13. doi: 10.2147/copd.s6643. Epub 2009 Sep 1. PMID 19750190
- [Result] Dougherty CM, Steele BG, Hunziker J. Testing an intervention to improve functional capability in advanced cardiopulmonary illness. J Cardiopulm Rehabil Prev. 2011 Jan-Feb;31(1):35-41. doi: 10.1097/HCR.0b013e3181f1fd77. PMID 20861749
- [Derived] Nguyen HQ, Steele BG, Dougherty CM, Burr RL. Physical activity patterns of patients with cardiopulmonary illnesses. Arch Phys Med Rehabil. 2012 Dec;93(12):2360-6. doi: 10.1016/j.apmr.2012.06.022. Epub 2012 Jul 5. PMID 22772084

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self-management | Usual Care
Started | 46 | 44
Completed | 42 | 38
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-management | Usual Care | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (10) | 66.4 (8) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Function Capability
Description: 6MWT-Six Minute Walk Test
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Self-management | Usual Care
Number analyzed (Participants) | 46 | 44
meters | 349 (146) | 338 (122)

2. Secondary Outcome: Quality of Life
Description: SF-36 PCS. Scale range 0-100, higher scores reflect higher quality of life. PCS=Physical Composite Score. These are not change scores.
Time Frame: 6 months
Population: These are not change scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-management | Usual Care
Number analyzed (Participants) | 46 | 44
units on a scale | 31 (8) | 38 (13)

ADVERSE EVENTS:
Arm/Group | Self-management | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes